CLINICAL TRIAL: NCT05694845
Title: A Clinical Study Experiences of Cholangiocarcinoma Patients To Identify Trial Attributes Affecting Completion Rates For Specific Demographic Groups
Brief Title: Evaluation of the Patient's Experience in Medical Studies for Cholangiocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82275501
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-01

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main reason for conducting this research is to gain a better understanding of why some people with cholangiocarcinoma are not able to participate in or complete clinical trials. Historically, certain groups of people have been more likely to participate in clinical trials, but there hasn't been much research to understand why this is the case.

The goal is to find out which aspects of a clinical trial may make it more difficult for patients to take part or see it through. The data will be evaluated through different demographic lenses and identify trends that could help improve the experience of future cholangiocarcinoma patients during clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Participant has a diagnosis of Cholangiocarcinoma
* Patient has self-identified as planning to enroll in an interventional Cholangiocarcinoma clinical trial
* Patient must provide written informed consent

Exclusion Criteria:

* No diagnosis of Cholangiocarcinoma confirmed
* Inability to perform regular electronic reporting
* Women who are pregnant, intend to become pregnant, or are lactating
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cholangiocarcinoma patients who are actively considering involvement in an observational clinical trial, but have not yet completed enrollment and registration.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a Cholangiocarcinoma Clinical Study. | 3 months
Number of Cholangiocarcinoma patients who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blechacz B, Komuta M, Roskams T, Gores GJ. Clinical diagnosis and staging of cholangiocarcinoma. Nat Rev Gastroenterol Hepatol. 2011 Aug 2;8(9):512-22. doi: 10.1038/nrgastro.2011.131. PMID 21808282
- [Background] Garcia-Pardo M, Ortega L, Fernandez-Acenero MJ, Garcia Alfonso P, Martin M, Munoz AJ. Molecular Profiling and Targeted Therapy in Cholangiocarcinoma: An Observational, Retrospective Multicenter Study. J Gastrointest Cancer. 2021 Jun;52(2):814-818. doi: 10.1007/s12029-021-00622-0. Epub 2021 Mar 8. PMID 33683644
- [Background] Ilyas SI, Khan SA, Hallemeier CL, Kelley RK, Gores GJ. Cholangiocarcinoma - evolving concepts and therapeutic strategies. Nat Rev Clin Oncol. 2018 Feb;15(2):95-111. doi: 10.1038/nrclinonc.2017.157. Epub 2017 Oct 10. PMID 28994423

DOCUMENTS (1):
  • Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT05694845/ICF_000.pdf